CLINICAL TRIAL: NCT01037764
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Acute Lymphoblastic Leukemia in Remission Using HLA-matched Sibling Donors, HLA-matched Unrelated Donors, or HLA-mismatched Familial Donors-A Phase 2 Study
Brief Title: Donor-specific Allogeneic Hematopoietic Cell Transplantation for Acute Lymphoblastic Leukemia (ALL)
Acronym: AHCTALL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI resigned the institute, and the rest investigators at the institute decided to terminate the study.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae-Young Kim, Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-ALLO-036
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Acute Lymphoid Leukemia
Keywords: acute lymphoid leukemia; primary complete remission; secondary complete remission; postremission therapy; allogeneic hematopoietic cell transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- alloHCT (Experimental): alloHCT arm: For HLA-matched sibling HCT, if a patient is 55 years old or less and without co-morbidity, the patient will receive Bu-Cy conditioning therapy and be transplanted with bone marrow cells. Patients who are older than 55 years or with co-morbidity will receive Bu-Flu-ATG conditioning and be transplanted with mobilized peripheral blood hematopoietic cells. For HLA-matched unrelated donor or HLA-mismatched familial donor HCT, the patient will receive Bu-Flu-ATG conditioning and well be transplanted with mobilized peripheral blood hematopoietic cells.
  Interventions: Procedure: alloHCT

INTERVENTIONS:
Procedure: alloHCT — [ alloHCT arm ] Bu-Cy conditioning; Busulfan (Bu) 3.2 mg/kg*/day iv daily on days -7 and -4. Cyclophosphamide (Cy) 60 mg/kg* in D5W 200 mL iv over 1-2 hours daily on days -3 and -2.
  BuFluATG conditioning; Bu 3.2 mg/kg*/day iv daily on days -7 and -6. Fludarabine (Flu) 30 mg/m2/day in D5W 100 ml iv over 30 minutes starting at 4 pm daily on days -7, -6, -5, -4, -3, and -2.
  Anti-thymocyte globulin (ATG, Thymoglobulin, Genzyme Transplant, Cambridge, MA, USA) 1.5 mg/kg/day (for HLA-matched sibling HCT) or 3.0 mg/kg/day (for HLA-matched unrelated donor HCT or HLA-mismatched familial donor HCT) in N/S 500-800 ml (less than 4 mg/ml) iv over 4 hours starting at 8 am daily on days , -3, -2 and -1.
  Other Names: allogeneic hematopoietic stem cell transplantation

SUMMARY:
[Study Objectives]

* To evaluate the efficacy of allogeneic hematopoietic cell transplantation (HCT) in patients with acute lymphoblastic leukemia (ALL) in the first or second complete remission (CR). The efficacy of the treatment will be measured in terms of the frequency of relapse and duration of remission (the primary endpoints).
* The secondary end points of the study include; engraftment, donor chimerism, secondary graft failure, acute and chronic graft-versus-host disease (GVHD), immune recovery, infections, transplantation-related mortality, leukemia free survival, and overall survival.

DETAILED DESCRIPTION:
1.0 STUDY OBJECTIVES

1.1. To evaluate the efficacy of allogeneic hematopoietic cell transplantation (HCT) in patients with acute lymphoblastic leukemia (ALL) either who have achieved complete remission (CR) after induction chemotherapy or who experienced recurrent leukemia then achieved second CR after salvage chemotherapy. The efficacy of the treatment will be measured in terms of the frequency of relapse after HCT and the duration of remission (the primary endpoints).

1.2. The secondary end points of the study include; engraftment (absolute neutrophil count over 500/㎕, unsupported platelet count over 20,000/㎕), donor chimerism at 2 and 4 weeks after HCT, secondary graft failure, acute and chronic graft-versus-host disease (GVHD), lymphocyte subset recovery at 1, 2, 3, 6, and 12 months, cytomegalovirus (CMV) reactivation/CMV disease, Epstein-Barr virus (EBV) reactivation/post-transplant lymphoproliferative disorder, transplantation-related mortality (100 day, 1 year), leukemia free survival, and overall survival.

1. 3. The hematopoietic cell donors in the study will include; HLA-matched sibling donors, HLA-matched unrelated donors, and HLA-mismatched family members, so that the majority of patients who achieve CR after induction or salvage chemotherapy will undergo allogeneic HCT as a part of consolidation therapy.

2.0 BACKGROUND INFORMATION

2.1. ALL is a malignant disorder characterized by the rapid proliferation of immature lymphocytes, which results in the accumulation and infiltration of neoplastic lymphocytes in the blood/bone marrow and other tissues. Allogeneic HCT is a curative therapeutic modality for a significant proportion of patients with ALL. Allogeneic HCT from HLA-matched sibling donors can produced long-term leukemia free survival in patients with ALL in high-risk first CR or second CR.(1) In adults with standard-risk ALL, the greatest benefit is achieved from a matched sibling allogeneic transplantation when compared to autologous transplantation or consolidation/maintenance therapy in the first CR status.(2)

2.2. Wider application of allogeneic HCT in patients with ALL, however, is impeded by limited donor availability. Less than a third of patients who need allogeneic HCT will have a HLA-matched sibling who can donate hematopoietic cells. For those patients who do not have an HLA-matched donor in the family, provided that they do not carry rare or private HLA-haplotype, HLA-matched unrelated donor can be found.(3) The chance of finding a willing unrelated donor in Korea is about 50%. On the other hand, nearly all patients who are in the need of allogeneic HCT have at least one HLA-haploidentical familial member, who is most willing to give hematopoietic cells immediately, not only for the initial transplantation, but also for the subsequent additional donations, if those became necessary. Early attempts to transplant allogeneic hematopoietic cells across the barriers of HLA-haplotype difference was met with high frequencies of engraftment failure and severe graft-versus-host disease (GVHD).(4, 5) Depletion of donor T cells from the graft before HCT decreased the frequency and severity of GVHD. However, it resulted in increased graft failure, delayed immune reconstitution, and increased fatal infections.(6-8) Further efforts to improve the outcomes of HLA-mismatched familial donor HCT included use of polyclonal(9, 10) or monoclonal antibodies(11, 12) against T cell as a part of conditioning regimen (in vivo-T cell depletion) and incorporation of the concept of feto-maternal immune tolerance in the donor selection process among several available HLA-haploidentical family members.(13)

2.3. In addition to aforementioned approaches, use of RIC in the setting of HLA-mismatched familial donor HCT has been explored. Various RIC regimens, utilizing total body irradiation (TBI),(14, 15) busulfan,(16, 17) or melphalan,(18) along with fludarabine, have been shown to be effective in achieving successful engraftment with less transplantation-related mortality (TRM), especially in elderly patients and in patients with organ dysfunctions, in the setting of HLA-matched donor HCT. These findings showed that under adequate immunosuppression, but not necessarily myeloablation, of the patients, donor hematopoietic cells can engraft and complete donor hematopoietic chimerism can be achieved. There are data that suggest the same principle may be extended to HLA-mismatched HCT settings as well. Successful engraftment of allogeneic hematopoietic cells across HLA-haplotype difference has been well-documented after RIC in animal models,(19-21) and in infants with severe combined immunodeficiency syndrome.(22, 23) In adult patient with hematologic malignancies, several studies involving small number of patients showed feasibility of successful engraftment of hematopoietic cell graft from HLA-haploidentical familial donor after RIC.(24-27)

2.4. Data generated in our hospital enhance the evidence of feasibility of hematopoietic engraftment across the HLA-haplotype barrier in adult patients after RIC.(28) Between April 2004 and February 2008, 31 patients (including 21 patients with acute leukemia) underwent HLA-haploidentical HCT after RIC of busulfan, fludarabine, and ATG and all 28 evaluable patients achieved engraftment with absolute lymphocyte count (ANC) over 500/㎕ on median day 16.5. As early as 2 weeks after HCT, 22 of 24 evaluated patients showed complete donor chimerism of 95% or over. None of the patients in the study experienced secondary graft failure. While achieving consistent and durable donor cell engraftment, the cumulative incidences of grades 2-4 acute and chronic GVHD were 19%, and 20%, respectively.

2.5. Between May 2008 and May 2009, 31 additional patients with acute leukemia were treated with HLA-mismatched HCT using the same treatment strategy as in the aforementioned study. As such, the data of 52 patients are now available. There were 24 male and 28 female with median age of 39.5 years (range, 16-70). Thirty-seven patients had AML, 13 ALL, and 2 acute mixed lineage leukemia. Ten patients were in first CR status, 15 in second or third CR status, and 27 had refractory disease. The donors were either offsprings (n=23), mothers (n=16), or siblings (n=13) of the patients and their median age was 37 years (range, 3-68). The conditioning regimen for HCT included busulfan in reduced-dose, fludarabine, and antithymocyte globulin. GVHD prophylaxis was given with cyclosporine and methotrexate. Other than 4 patients who experienced leukemia progression within 30 days of HCT or died early, all the rest 48 patients achieved donor cell engraftment with absolute neutrophil count (ANC) >500/㎕ on median 14.5 days (range, 10-27). One patient experienced secondary graft failure subsequently. Cumulative incidence rates for acute GVHD grade 2-4 and chronic GVHD were 10% (95% CI, 4%-23%) and 33% (95% CI, 22%-51%), respectively. Cumulative incidence rates of leukemia progression/recurrence were 13%, 41%, and 77% for patients in CR1, CR2-3, and refractory leukemia at the time of HCT. In all, five patients in the series died without leukemia progression/recurrence giving transplantation-related mortality (TRM) rate of 12% (95% CI, 5%-29%). Kaplan-Meier event-free survival and overall survival rates were 44% and 50% for patients in CR1 at HCT, 40% and 23% for patients in CR2-3, and 10% and 15% for patients with refractory leukemia. These results showed that HCT from an HLA-mismatched family member can be performed in patients with acute leukemia successfully without increased GVHD or TRM.

2.6. In our current prospective study, we try to integrate HLA-mismatched HCT in overall care of patients with ALL in the first or second CR. In the past, those patients without an HLA-matched donor in the family or unrelated donor registry were not offered allogeneic HCT. The outcomes of HCT will be analyzed according to several clinical variables such as patient, disease, and donor characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ALL who achieve CR after induction chemotherapy.
* Patients with recurrent ALL that went into second CR after salvage chemotherapy, except those who had undergone allogeneic HCT previously.
* Patients should be 15 years of age or more, and 75 years of age or less.
* The performance status of the patients should be 70 or over by Karnofsky performance scale.
* Patients should have adequate hepatic function (bilirubin less than 2.0 mg/dl, AST less than three times the upper normal limit).
* Patients must have adequate renal function (creatinine less than 2.0 mg/dl).
* Patients must have adequate cardiac function (ejection fraction > 40% on MUGA scan).
* Patients must sign informed consent.

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of relapse | 3 years

SECONDARY OUTCOMES:
leukemia free survival | 3 years
engraftment rate | 100 days
donor chimerism | 1year, 2year, 3year
secondary graft failure rate | 100days, 1year
Incidence & severity of acute GVHD | 100 days
incidence and severity of chronic GVHD | 1year, 2year, 3year
degree of immune recovery | 6 months, 1year
cumulative incidence and severity of infection | 3years
transplantation-related mortality rate | 3 years
overall survival rate & median survival time | 3 years
duration of remission | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Young Kim, M.D. & PhD, Principal Investigator — Asan Medical Center; Kyoo-Hyung Lee, M.D. & PhD., Study Chair — Asan Medical Center; Je-Hwan Lee, M.D. & PhD., Study Director — Asan Medical Center; Jung-Hee Lee, M.D. & PhD., Study Director — Asan Medical Center; Young-Don Joo, MD, PhD, Study Director — Inje University Haeundae Paik Hospital
Locations (2):
- South Korea (2):
  - Inje University Haeundae Paik Hospital, Pusan
  - Asan Medical Center, Seoul

REFERENCES:
- [Background] Jamieson CH, Amylon MD, Wong RM, Blume KG. Allogeneic hematopoietic cell transplantation for patients with high-risk acute lymphoblastic leukemia in first or second complete remission using fractionated total-body irradiation and high-dose etoposide: a 15-year experience. Exp Hematol. 2003 Oct;31(10):981-6. doi: 10.1016/s0301-472x(03)00231-5. PMID 14550815
- [Background] Goldstone AH, Richards SM, Lazarus HM, Tallman MS, Buck G, Fielding AK, Burnett AK, Chopra R, Wiernik PH, Foroni L, Paietta E, Litzow MR, Marks DI, Durrant J, McMillan A, Franklin IM, Luger S, Ciobanu N, Rowe JM. In adults with standard-risk acute lymphoblastic leukemia, the greatest benefit is achieved from a matched sibling allogeneic transplantation in first complete remission, and an autologous transplantation is less effective than conventional consolidation/maintenance chemotherapy in all patients: final results of the International ALL Trial (MRC UKALL XII/ECOG E2993). Blood. 2008 Feb 15;111(4):1827-33. doi: 10.1182/blood-2007-10-116582. Epub 2007 Nov 29. PMID 18048644
- [Background] Barker JN, Krepski TP, DeFor TE, Davies SM, Wagner JE, Weisdorf DJ. Searching for unrelated donor hematopoietic stem cells: availability and speed of umbilical cord blood versus bone marrow. Biol Blood Marrow Transplant. 2002;8(5):257-60. doi: 10.1053/bbmt.2002.v8.pm12064362.
- [Background] Powles RL, Morgenstern GR, Kay HE, McElwain TJ, Clink HM, Dady PJ, Barrett A, Jameson B, Depledge MH, Watson JG, Sloane J, Leigh M, Lumley H, Hedley D, Lawler SD, Filshie J, Robinson B. Mismatched family donors for bone-marrow transplantation as treatment for acute leukaemia. Lancet. 1983 Mar 19;1(8325):612-5. doi: 10.1016/s0140-6736(83)91793-2. PMID 6131300
- [Background] Beatty PG, Clift RA, Mickelson EM, Nisperos BB, Flournoy N, Martin PJ, Sanders JE, Stewart P, Buckner CD, Storb R, et al. Marrow transplantation from related donors other than HLA-identical siblings. N Engl J Med. 1985 Sep 26;313(13):765-71. doi: 10.1056/NEJM198509263131301. PMID 3897863
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Henslee-Downey PJ, Abhyankar SH, Parrish RS, Pati AR, Godder KT, Neglia WJ, Goon-Johnson KS, Geier SS, Lee CG, Gee AP. Use of partially mismatched related donors extends access to allogeneic marrow transplant. Blood. 1997 May 15;89(10):3864-72. PMID 9160695
- [Background] Lacerda JF, Martins C, Carmo JA, Lourenco F, Juncal C, Rodrigues A, Vilalobos I, Moura MC, Ligeiro D, Martinho A, Lacerda JM. Haploidentical stem cell transplantation with purified CD34 cells after a chemotherapy-alone conditioning regimen. Biol Blood Marrow Transplant. 2003 Oct;9(10):633-42. doi: 10.1016/s1083-8791(03)00263-5. PMID 14569559
- [Background] Huang XJ, Liu DH, Liu KY, Xu LP, Chen H, Han W, Chen YH, Wang JZ, Gao ZY, Zhang YC, Jiang Q, Shi HX, Lu DP. Haploidentical hematopoietic stem cell transplantation without in vitro T-cell depletion for the treatment of hematological malignancies. Bone Marrow Transplant. 2006 Aug;38(4):291-7. doi: 10.1038/sj.bmt.1705445. PMID 16883312
- [Background] Kanda Y, Oshima K, Asano-Mori Y, Kandabashi K, Nakagawa M, Sakata-Yanagimoto M, Izutsu K, Hangaishi A, Tsujino S, Ogawa S, Motokura T, Chiba S, Hirai H. In vivo alemtuzumab enables haploidentical human leukocyte antigen-mismatched hematopoietic stem-cell transplantation without ex vivo graft manipulation. Transplantation. 2005 May 27;79(10):1351-7. doi: 10.1097/01.tp.0000158718.49286.14. PMID 15912103
- [Background] DiJerome L. The nursing case management computerized system: meeting the challenge of health care delivery through technology. Comput Nurs. 1992 Nov-Dec;10(6):250-8. PMID 1458364
- [Background] Ichinohe T, Uchiyama T, Shimazaki C, Matsuo K, Tamaki S, Hino M, Watanabe A, Hamaguchi M, Adachi S, Gondo H, Uoshima N, Yoshihara T, Hatanaka K, Fujii H, Kawa K, Kawanishi K, Oka K, Kimura H, Itoh M, Inukai T, Maruya E, Saji H, Kodera Y; Japanese Collaborative Study Group for NIMA-Complementary Haploidentical Stem Cell Transplantation. Feasibility of HLA-haploidentical hematopoietic stem cell transplantation between noninherited maternal antigen (NIMA)-mismatched family members linked with long-term fetomaternal microchimerism. Blood. 2004 Dec 1;104(12):3821-8. doi: 10.1182/blood-2004-03-1212. Epub 2004 Jul 27. PMID 15280193
- [Background] McSweeney PA, Niederwieser D, Shizuru JA, Sandmaier BM, Molina AJ, Maloney DG, Chauncey TR, Gooley TA, Hegenbart U, Nash RA, Radich J, Wagner JL, Minor S, Appelbaum FR, Bensinger WI, Bryant E, Flowers ME, Georges GE, Grumet FC, Kiem HP, Torok-Storb B, Yu C, Blume KG, Storb RF. Hematopoietic cell transplantation in older patients with hematologic malignancies: replacing high-dose cytotoxic therapy with graft-versus-tumor effects. Blood. 2001 Jun 1;97(11):3390-400. doi: 10.1182/blood.v97.11.3390. PMID 11369628
- [Background] Hegenbart U, Niederwieser D, Sandmaier BM, Maris MB, Shizuru JA, Greinix H, Cordonnier C, Rio B, Gratwohl A, Lange T, Al-Ali H, Storer B, Maloney D, McSweeney P, Chauncey T, Agura E, Bruno B, Maziarz RT, Petersen F, Storb R. Treatment for acute myelogenous leukemia by low-dose, total-body, irradiation-based conditioning and hematopoietic cell transplantation from related and unrelated donors. J Clin Oncol. 2006 Jan 20;24(3):444-53. doi: 10.1200/JCO.2005.03.1765. Epub 2005 Dec 12. PMID 16344316
- [Background] Lee KH, Lee JH, Lee JH, Kim WK, Chi HS, Lee JS. Non-myeloablative conditioning regimen of fludarabine, busulfan, anti-thymocyte globulin, and methylprednisolone for allogeneic peripheral blood hematopoietic cell transplantation. Haematologica. 2001 Sep;86(9):999-1001. No abstract available. PMID 11532635
- [Background] Alyea EP, Kim HT, Ho V, Cutler C, Gribben J, DeAngelo DJ, Lee SJ, Windawi S, Ritz J, Stone RM, Antin JH, Soiffer RJ. Comparative outcome of nonmyeloablative and myeloablative allogeneic hematopoietic cell transplantation for patients older than 50 years of age. Blood. 2005 Feb 15;105(4):1810-4. doi: 10.1182/blood-2004-05-1947. Epub 2004 Sep 30. PMID 15459007
- [Background] Giralt S, Thall PF, Khouri I, Wang X, Braunschweig I, Ippolitti C, Claxton D, Donato M, Bruton J, Cohen A, Davis M, Andersson BS, Anderlini P, Gajewski J, Kornblau S, Andreeff M, Przepiorka D, Ueno NT, Molldrem J, Champlin R. Melphalan and purine analog-containing preparative regimens: reduced-intensity conditioning for patients with hematologic malignancies undergoing allogeneic progenitor cell transplantation. Blood. 2001 Feb 1;97(3):631-7. doi: 10.1182/blood.v97.3.631. PMID 11157478
- [Background] Cina RA, Wikiel KJ, Lee PW, Cameron AM, Hettiarachy S, Rowland H, Goodrich J, Colby C, Spitzer TR, Neville DM Jr, Huang CA. Stable multilineage chimerism without graft versus host disease following nonmyeloablative haploidentical hematopoietic cell transplantation. Transplantation. 2006 Jun 27;81(12):1677-85. doi: 10.1097/01.tp.0000226061.59196.84. PMID 16794534
- [Background] Fukuda T, Kerbauy FR, Gooley T, Santos EB, Storb R, Sandmaier BM. Dog leukocyte antigen-haploidentical stem cell allografts after anti-CD44 therapy and nonmyeloablative conditioning in a preclinical canine model. Transplantation. 2006 Aug 15;82(3):332-9. doi: 10.1097/01.tp.0000228908.10775.b0. PMID 16906030
- [Background] Vanclee A, Lutgens LC, Oving EB, Deutz NE, Gijbels MJ, Schouten HC, Bos GM. Keratinocyte growth factor ameliorates acute graft-versus-host disease in a novel nonmyeloablative haploidentical transplantation model. Bone Marrow Transplant. 2005 Nov;36(10):907-15. doi: 10.1038/sj.bmt.1705157. PMID 16151417
- [Background] Fischer A, Durandy A, de Villartay JP, Vilmer E, Le Deist F, Gerota I, Griscelli C. HLA-haploidentical bone marrow transplantation for severe combined immunodeficiency using E rosette fractionation and cyclosporine. Blood. 1986 Feb;67(2):444-9. PMID 3510681
- [Background] Haddad E, Landais P, Friedrich W, Gerritsen B, Cavazzana-Calvo M, Morgan G, Bertrand Y, Fasth A, Porta F, Cant A, Espanol T, Muller S, Veys P, Vossen J, Fischer A. Long-term immune reconstitution and outcome after HLA-nonidentical T-cell-depleted bone marrow transplantation for severe combined immunodeficiency: a European retrospective study of 116 patients. Blood. 1998 May 15;91(10):3646-53. PMID 9573000
- [Background] Sykes M, Preffer F, McAfee S, Saidman SL, Weymouth D, Andrews DM, Colby C, Sackstein R, Sachs DH, Spitzer TR. Mixed lymphohaemopoietic chimerism and graft-versus-lymphoma effects after non-myeloablative therapy and HLA-mismatched bone-marrow transplantation. Lancet. 1999 May 22;353(9166):1755-9. doi: 10.1016/S0140-6736(98)11135-2. PMID 10347989
- [Background] Spitzer TR, McAfee SL, Dey BR, Colby C, Hope J, Grossberg H, Preffer F, Shaffer J, Alexander SI, Sachs DH, Sykes M. Nonmyeloablative haploidentical stem-cell transplantation using anti-CD2 monoclonal antibody (MEDI-507)-based conditioning for refractory hematologic malignancies. Transplantation. 2003 May 27;75(10):1748-51. doi: 10.1097/01.TP.0000064211.23536.AD. PMID 12777868
- [Background] O'Donnell PV, Luznik L, Jones RJ, Vogelsang GB, Leffell MS, Phelps M, Rhubart P, Cowan K, Piantados S, Fuchs EJ. Nonmyeloablative bone marrow transplantation from partially HLA-mismatched related donors using posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2002;8(7):377-86. doi: 10.1053/bbmt.2002.v8.pm12171484.
- [Background] Tamaki H, Ikegame K, Kawakami M, Fujioka T, Tsuboi A, Oji Y, Oka Y, Sugiyama H, Kawase I, Ogawa H. Successful engraftment of HLA-haploidentical related transplants using nonmyeloablative conditioning with fludarabine, busulfan and anti-T-lymphocyte globulin. Leukemia. 2003 Oct;17(10):2052-4. doi: 10.1038/sj.leu.2403092. No abstract available. PMID 14513058
- [Background] Byrd JC, Mrozek K, Dodge RK, Carroll AJ, Edwards CG, Arthur DC, Pettenati MJ, Patil SR, Rao KW, Watson MS, Koduru PR, Moore JO, Stone RM, Mayer RJ, Feldman EJ, Davey FR, Schiffer CA, Larson RA, Bloomfield CD; Cancer and Leukemia Group B (CALGB 8461). Pretreatment cytogenetic abnormalities are predictive of induction success, cumulative incidence of relapse, and overall survival in adult patients with de novo acute myeloid leukemia: results from Cancer and Leukemia Group B (CALGB 8461). Blood. 2002 Dec 15;100(13):4325-36. doi: 10.1182/blood-2002-03-0772. Epub 2002 Aug 1. PMID 12393746
- [Background] Lee KH, Lee JH, Lee JH, Kim DY, Kim SH, Shin HJ, Lee YS, Kang YA, Seol M, Ryu SG. Hematopoietic cell transplantation from an HLA-mismatched familial donor is feasible without ex vivo-T cell depletion after reduced-intensity conditioning with busulfan, fludarabine, and antithymocyte globulin. Biol Blood Marrow Transplant. 2009 Jan;15(1):61-72. doi: 10.1016/j.bbmt.2008.10.025. PMID 19135944
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616